CLINICAL TRIAL: NCT03529552
Title: Short-, Medium- and Long-term (up to 3 Years) Evaluation After Reconstruction of the Anterior Cruciate Ligament of the Knee Using the Bioresorbable Interference Screw (SMS): Resorbability, Per- and Post-operative Complications and Articular Functional Recovery.
Brief Title: Evaluation After Reconstruction of the Anterior Cruciate Ligament of the Knee Using the Bioresorbable Interference Screw (SMS): Resorbability, Per- and Post-operative Complications and Articular Functional Recovery.
Acronym: BIORELICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Dm production has been stopped
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Dedienne Sante S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDIL/2017/PM-01
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with anterior cruciate ligament rupture (Experimental)
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction

INTERVENTIONS:
Procedure: Anterior Cruciate Ligament Reconstruction — Placement of an SMS bioresorbable interference screw (DEDIENNE Santé)

SUMMARY:
The investigators will evaluate the benefit of a new bioresorbable screw for repair of anterior cruciate ligament over 3 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient is available for at least 3 years of follow-up
* The patient requires ligamentoplasty pour rupture of anterior cruciate ligament confirmed by MRI with or without meniscal lesions as scheduled surgery

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breast-feeding
* The patient has a contra-indication (or a medically-incompatible association) for the treatment, including MRI
* Revision surgery
* Simultaneous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
In situ degradation of screw | Year 3
  Assessed on T1 and proton density fat saturation MRI

SECONDARY OUTCOMES:
Knee stiffness | Day -1
  Articular amplitude test
Knee stiffness | Day 0
  Articular amplitude test
Knee stiffness | Week 6
  Articular amplitude test
Knee stiffness | Month 3
  Articular amplitude test
Knee stiffness | Month 8
  Articular amplitude test
Knee stiffness | Year 1
  Articular amplitude test
Knee stiffness | Year 2
  Articular amplitude test
Knee stiffness | Year 3
  Articular amplitude test
Knee mobility | Day -1
  Anterior pull test
Knee mobility | Day 0
  Anterior pull test
Knee mobility | Week 6
  Anterior pull test
Knee mobility | Month 3
  Anterior pull test
Knee mobility | Month 8
  Anterior pull test
Knee mobility | Year 1
  Anterior pull test
Knee mobility | Year 2
  Anterior pull test
Knee mobility | Year 3
  Anterior pull test
Lateral pivot shift of knee | Day -1
  MacIntosh test
Lateral pivot shift of knee | Day 0
  MacIntosh test
Lateral pivot shift of knee | Week 6
  MacIntosh test
Lateral pivot shift of knee | Month 3
  MacIntosh test
Lateral pivot shift of knee | Month 8
  MacIntosh test
Lateral pivot shift of knee | Year 1
  MacIntosh test
Lateral pivot shift of knee | Year 2
  MacIntosh test
Lateral pivot shift of knee | Year 3
  MacIntosh test
Impact of knee pain on daily life | Day -1
  Lysholm Knee Scoring Scale
Impact of knee pain on daily life | Day 0
  Lysholm Knee Scoring Scale
Impact of knee pain on daily life | Week 6
  Lysholm Knee Scoring Scale
Impact of knee pain on daily life | Month 3
  Lysholm Knee Scoring Scale
Impact of knee pain on daily life | Month 8
  Lysholm Knee Scoring Scale
Impact of knee pain on daily life | year 1
  Lysholm Knee Scoring Scale
Impact of knee pain on daily life | Year 2
  Lysholm Knee Scoring Scale
Impact of knee pain on daily life | Year 3
  Lysholm Knee Scoring Scale
Patient-reported knee problems | Day -1
  International Knee Documentation Committee Questionnaire
Patient-reported knee problems | Day 0
  International Knee Documentation Committee Questionnaire
Patient-reported knee problems | Week 6
  International Knee Documentation Committee Questionnaire
Patient-reported knee problems | Month 3
  International Knee Documentation Committee Questionnaire
Patient-reported knee problems | Month 8
  International Knee Documentation Committee Questionnaire
Patient-reported knee problems | Year 1
  International Knee Documentation Committee Questionnaire
Patient-reported knee problems | Year 2
  International Knee Documentation Committee Questionnaire
Patient-reported knee problems | Year 3
  International Knee Documentation Committee Questionnaire
Knee laxity | Day -1
  KT-1000 measurement
Knee laxity | Day 0
  KT-1000 measurement
Knee laxity | Week 6
  KT-1000 measurement
Knee laxity | Month 3
  KT-1000 measurement
Knee laxity | Month 8
  KT-1000 measurement
Knee laxity | Year 1
  KT-1000 measurement
Knee laxity | Year 2
  KT-1000 measurement
Knee laxity | Year 3
  KT-1000 measurement
Passive accessory movement of knee | Day -1
  Lachman test
Passive accessory movement of knee | Day 0
  Lachman test
Passive accessory movement of knee | Week 6
  Lachman test
Passive accessory movement of knee | Month 3
  Lachman test
Passive accessory movement of knee | Month 8
  Lachman test
Passive accessory movement of knee | Year 1
  Lachman test
Passive accessory movement of knee | Year 2
  Lachman test
Passive accessory movement of knee | Year 3
  Lachman test
Anterior cruciate ligament and posterior capsule integrity | Day -1
  Pivot-shift test
Anterior cruciate ligament and posterior capsule integrity | Day 0
  Pivot-shift test
Anterior cruciate ligament and posterior capsule integrity | Week 6
  Pivot-shift test
Anterior cruciate ligament and posterior capsule integrity | Month 3
  Pivot-shift test
Anterior cruciate ligament and posterior capsule integrity | Month 8
  Pivot-shift test
Anterior cruciate ligament and posterior capsule integrity | Year 1
  Pivot-shift test
Anterior cruciate ligament and posterior capsule integrity | Year 2
  Pivot-shift test
Anterior cruciate ligament and posterior capsule integrity | Year 3
  Pivot-shift test
Post-operative complications | Year 3
  Undesirable events

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Marchand, MD, Principal Investigator — CHU Nimes
Locations (3):
- France (3):
  - Polyclinique Urbain V, Avignon
  - Centre Régina, Nice
  - CHU Nimes, Nîmes